CLINICAL TRIAL: NCT05418101
Title: A Phase 1, First-in-human, 2-part Study (part 1 is a Single Ascending Dose in Healthy Participants; Part 2 is a Multiple Ascending Dose Study in Participants with Autoimmune Disease) to Evaluate the Safety, PD and PK of VIS171
Brief Title: A Study to Evaluate the Safety, PK and PD of VIS171 in Participants (Healthy and with Autoimmune Disease)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Visterra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VIS171-101; 2021-006246-12 (EudraCT Number)
Record Dates: First submitted 2022-06-03; First posted 2022-06-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-04

CONDITIONS: Autoimmune Diseases
Keywords: Safety; Tolerability; Pharmacodynamics; Pharmacokinetics; Healthy participants
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: This phase 1 study has two parts. Part A is a randomized, double-blind, placebo controlled SAD assessment of SC VIS171 in healthy participants. Part B is an open-label, MAD basket assessment of SC VIS171 in participants with an autoimmune inflammatory disease
Masking Description: Part A will be double masked; Part B is open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Part A Cohort 1: Dose level 1 (Experimental): Participants will be randomized to SAD dose of VIS171 (or placebo).
  Interventions: Drug: VIS171; Drug: Placebo
- Part A Cohort 2: Dose level 2 (Experimental): Participants will be randomized to SAD dose of VIS171 (or placebo).
  Interventions: Drug: VIS171; Drug: Placebo
- Part A Cohort 3: Dose level 3 (Experimental): Participants will be randomized to SAD dose of VIS171 (or placebo).
  Interventions: Drug: VIS171; Drug: Placebo
- Part A Cohort 4: Dose level 4 (Experimental): Participants will be randomized to SAD dose of VIS171 (or placebo).
  Interventions: Drug: VIS171; Drug: Placebo
- Part A Cohort 5: Dose level 5 (Experimental): Participants will be randomized to SAD dose of VIS171 (or placebo).
  Interventions: Drug: VIS171; Drug: Placebo
- Part B Cohort 1: Dose level to be determined from SAD Cohort(s) data (Experimental): Participants will be randomized to MAD dose of VIS171.
  Interventions: Drug: VIS171
- Part B Cohort 2: Dose level to be determined from SAD Cohort(s) data (Experimental): Participants will be randomized to MAD dose of VIS171.
  Interventions: Drug: VIS171
- Part B Cohort 3: Dose level and regimen to be determined from prior MAD and SAD Cohort(s) (Experimental): Participants will be randomized to MAD dose of VIS171.
  Interventions: Drug: VIS171

INTERVENTIONS:
Drug: VIS171 — Participants will receive VIS171 via SC route of administration.
Drug: Placebo — Participants will receive Placebo via SC route of administration
  Arms: Part A Cohort 1: Dose level 1; Part A Cohort 2: Dose level 2; Part A Cohort 3: Dose level 3; Part A Cohort 4: Dose level 4; Part A Cohort 5: Dose level 5

SUMMARY:
This is a phase 1 study to evaluate the safety, tolerability, pharmacodynamics, and pharmacokinetics of VIS171 in healthy participants and in participants with autoimmune disease(s).

DETAILED DESCRIPTION:
This is a multicenter, 2-part combined Single ascending dose (SAD) and Multiple ascending dose (MAD) First-in-Human (FIH) study to investigate the safety, tolerability, pharmacodynamics (PD), and pharmacokinetics (PK) of subcutaneous (SC) VIS171 in healthy participants (Part A - SAD) and in participants with autoimmune inflammatory disease(s) (Part B - MAD).

Part A: Part A is a randomized, double-blind, placebo controlled SAD assessment of SC VIS171 in healthy participants. Up to 5 cohorts are planned, each comprising 8 participants (6 VIS171 and 2 placebo).

Part B: Part B is an open-label, MAD basket assessment of SC VIS171 in participants with autoimmune inflammatory disease(s). Two to 3 cohorts are planned, each comprising 12 participants.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for both Part A and Part B:

* Male or female participant between 18 and 55 years of age, inclusive, at the screening visit (Part A and Part B [participants with selected autoimmune diseases]) or between 18 and 75 years of age, inclusive, at the screening visit (Part B [participants with specific autoimmune disease]).
* Body mass index between 17 and 35 kg/m^2.
* Female participants will be nonpregnant, nonlactating, and either postmenopausal for at least 2 years or surgically sterile for at least 3 months.
* Male participants with female partners of childbearing potential must agree to use double barrier contraception or abstain from sex during the study and until 90 days following the last dose of study intervention.

Additional inclusion criterion for Part A:

- Healthy, as determined by prestudy medical evaluation (medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations).

Additional inclusion criteria for Part B (participants with specific autoimmune disease[s]):

* Diagnosis of a specified autoimmune disease based on standard criteria for the condition.
* Other criteria may apply depending on the autoimmune condition.

Exclusion Criteria:

Exclusion criteria for both Part A and Part B:

Prior and Concomitant Therapy

* Receipt of high dose corticosteroid therapy within 4 weeks prior to screening.
* Receipt of belimumab within 6 months prior to screening.
* History of treatment with rituximab or ocrelizumab (or other B cell-depleting agent) within 12 months prior to screening.
* History of cytotoxic medications within the preceding 12 months.
* Receipt of blood products within 6 months prior to screening.

Prior/Concurrent Clinical Study Experience:

* Receipt of any investigational product within 4 weeks or 5 half-lives of the respective product prior to signing of the ICF, whichever is greater.
* Currently participating in another clinical study of any investigational drug, device, or intervention.

Diagnostic Assessments

* Participants with uncontrolled hypertension (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg in any position) or symptomatic hypotension.
* Any chronic infectious disease.
* Participant with a positive urine drug or alcohol breath screen test result at screening.

Other Exclusions:

* Any participant who has a history of alcohol or drug/chemical abuse.
* Participant who has donated > 500 mL of blood within 60 days prior to the start of screening or any plasma within 7 days prior to baseline (Day -1).
* History of opportunistic infection requiring hospitalization or intravenous (IV) antimicrobial treatment within 1 year prior to randomization.
* History of major surgery within 12 weeks of screening or will require major surgery during the study.
* Clinically significant electrocardiographic abnormalities, at screening.
* A QT interval corrected for heart rate using Fridericia's correction (QTcF) > 450 msec for male participants or > 470 msec for female participants at screening.
* Participant has received an organ transplant.
* History of any significant cardiovascular disease or thrombotic episode.
* History of cancer, apart from: squamous or basal cell carcinoma of the skin that has been successfully treated; cervical cancer in situ that has been successfully treated.
* Coronavirus Disease 2019 (COVID-19): current symptoms of infection; diagnosis of COVID-19 in the 21 days prior to Screening; ongoing diagnosis of "Long-COVID" symptoms.
* Received a vaccination, other than COVID-19 vaccination, during the 30 days prior to administration of the first dose of study intervention. A COVID-19 vaccination cannot be received within 7 days prior to the first dose of study intervention and until 14 days after the last dose.

Additional exclusion criteria for Part A:

Medical Conditions

* Participant has a history or current evidence of a serious and/or unstable cardiovascular, respiratory, gastrointestinal, hematologic, autoimmune, blood dyscrasias or other medical disorder, including psychiatric disorders, cirrhosis, or malignancy.
* Participant has a history or presence of proteinuria, chronic kidney disease, disease requiring immunosuppressive therapy (including systemic steroids), or is considered to be immunosuppressed for any other reason.
* History of a previous severe allergic reaction with generalized urticaria; angioedema or anaphylaxis.
* Known immunodeficiency disorder.
* History of chronic infection or any infection requiring hospitalization or treatment with antivirals, antibiotics, or antifungal therapy within 30 days prior to administration of the study intervention.
* Alanine transaminase (ALT) or aspartate transaminase (AST) > 1.5 × the upper limit of normal (ULN).
* Total bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN is acceptable if total bilirubin is fractionated and direct bilirubin < 35%).
* Known hepatic or biliary abnormalities.

Additional exclusion criterion for Part A and Part B (participants with participants with specific autoimmune disease may apply depending upon the autoimmune condition).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Part A and Part B: Numbers of participants with treatment-emergent adverse events (TEAEs) | Part A: From screening up to Day 29; Part B: From screening up to Day 71

SECONDARY OUTCOMES:
Part A and Part B: Mean change from baseline in absolute number (cells/μL) for Treg, helper T cells, cytotoxic T cells and natural killer cells | Part A: From baseline up to Day 29; Part B: From baseline up to Day 71
Part A and Part B: Mean change from baseline in percentage for Treg, helper T cells, cytotoxic T cells and natural killer cells | Part A: From baseline up to Day 29; Part B: From baseline up to Day 71
Part A and Part B: Maximum (peak) plasma VIS171 concentration (Cmax) over time | Part A: From baseline up to Day 29; Part B: From baseline up to Day 71
Part A and Part B: Time of maximum (peak) plasma VIS171 concentration (tmax) | Part A: From baseline up to Day 29; Part B: From baseline up to Day 71
Part A: Area under the concentration-time curve from time zero to the last observable concentration (AUClast) of VIS171 | Part A: From baseline up to Day 29
Part A: Area under the concentration-time curve from time zero to infinity (AUC∞) for VIS171 concentration | Part A: From baseline up to Day 29
Part B: Area under the concentration-time curve over the dosing interval at steady-state (AUCtau) | Part B: From baseline up to Day 71
Part A and Part B: Number of participants with Anti-drug antibodies (ADA) positive for VIS171 | Part A: Day 1, 15, and 29; Part B: Day 1, 15, 29, 43, and 71

CONTACTS AND LOCATIONS:
Overall Officials: Asher Schachter, MD, Principal Investigator — Visterra, Inc.
Locations (10):
- Bulgaria (5):
  - UMHAT, Plovdiv
  - Ambulatory for Specialized Medical Help - skin and venereal diseases, Sofia
  - Comac Medical Ltd, Sofia
  - MBAL Sveta Sofia, Sofia
  - Diagnostic and Consultative Center Convex EOOD, Sofia
- Germany (2):
  - Universitaetsklinikum Bonn AöR, Bonn
  - Universitätsmedizin der Johannes-Gutenberg-Universität Mainz, Rheinland-Pfalz
- Clinical republican Hospital, Chisinau, Moldova
- Radboud University Medical Center, Gelderland, Netherlands
- New Zealand Clinical Research, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No